CLINICAL TRIAL: NCT07346261
Title: Impact of Digital High-Intensity Respiratory Muscle Training on Ventilatory Function and Functional Capacity in Patients With COPD
Brief Title: Digital High-Intensity Respiratory Muscle Training on COPD Patients
Acronym: COPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar Waly, principal investigator MSc candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/006187
Record Dates: First submitted 2026-01-15; First posted 2026-01-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A (study group) (Experimental): 30 patient who will receive high-intensity respiratory training with the digital Sonmol Respiratory Muscle Trainer for 15 to 20 Minutes, in addition to a conventional pulmonary rehabilitation program for 25 to 30 Minutes, with a total duration of 50 to 60 minutes for each session.
  , 3 sessions/week, for 8 weeks.
  Interventions: Device: Digital Sonmol Respiratory Muscle Trainer; Other: conventional respiratory rehabilitation
- Group B (control group) (Experimental): 30 patient who will receive the conventional pulmonary rehabilitation program for 25 to 30 minutes for each session, 3 sessions / week, for 8 weeks.
  Interventions: Other: conventional respiratory rehabilitation

INTERVENTIONS:
Device: Digital Sonmol Respiratory Muscle Trainer — The patient will be asked to inhale deeply and forcefully for approximately two to three seconds and have a pause of slightly under a second. Then exhale out of the device and rest for 30 to 60 seconds and will be done for 2 sets of ten breaths, two times per day, for eight weeks The resistance will increase about 10 % to 15 % every week according to patient status in addition to a conventional respiratory rehabilitation program for 25 to 30 Minutes, with a total duration of 50 to 60 minutes for each session.
  Arms: Group A (study group)
Other: conventional respiratory rehabilitation — The patients will receive conventional respiratory Rehabilitation in the form of Diaphragmatic breathing exercise for 5 to 10 minutes and Localized Breathing for lower, middle, and upper segments for 10 to 15 minutes, total session time 25 to 30 minutes for two to four sessions daily for 3 days/ week for 8 weeks

SUMMARY:
The goal of this Randomize control trail is to determine the effect of Digital High-Intensity Respiratory Muscle Training on ventilatory Function and Functional Capacity in Patients with COPD It will also learn about the safety and tolerability of this digital training program.

The main questions it aims to answer are: Does digital high-intensity respiratory muscle training improve inspiratory and expiratory muscle strength (MIP and MEP)? ,Does it improve functional exercise capacity (6-minute walk distance) and lung function (FEV₁, FVC, FEV₁/FVC)?

DETAILED DESCRIPTION:
This single-blinded randomized controlled trial is to determine effect of Digital High-intensity Respiratory Muscle Training delivered through the Sonmol electronic respiratory muscle trainer on ventilatory function and functional capacity in patients with chronic obstructive pulmonary diseases (COPD)

It articulates the clinical rationale by explaining how airflow limitation is caused by COPD and chest hyperinflation, or dysfunction of respiratory muscles, and describes why specific, intense exercise training of muscles of inspiration or expiration may correct or prevent these conditions.

This trial within current evidence supporting respiratory-muscle training and highlights the potential advantages of digital delivery-real-time feedback, adjustable resistance, gamification, and remote monitoring-to boost adherence and training specificity in a rehabilitation context.

The study compares digital high-intensity respiratory muscle training plus conventional pulmonary rehabilitation to conventional pulmonary rehabilitation alone to see if the digital training provides additional benefits.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of chronic obstructive pulmonary disease (COPD), moderate to severe (GOLD stage II-IV)
2. FEV₁ > 80% of predicted.
3. Age 50-65 years.
4. Able to perform high-intensity respiratory muscle training (MIP and MEP ≥ device threshold).
5. Clinically stable with no acute exacerbations.

Exclusion Criteria:

1. Severe comorbidities (e.g., coronary heart disease, arterial aneurysm, severe hepatic or renal dysfunction, uncontrolled hypertension).
2. Unstable medical conditions or other respiratory diseases that could cause or contribute to breathlessness (e.g., asthma, pneumonia, bronchiectasis, tuberculosis, interstitial lung disease).
3. Mental illness, deafness, limb activity disorder, or any condition causing inability to cooperate with procedures.
4. Cognitive impairment or psychiatric illness that affects cooperation.
5. Participation in another clinical trial or intervention within the last 3 months.
6. Current use of any other respiratory muscle training device or app.

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Ventilatory function measures (FVC, FEV1, and FEV1/FVC) | twice, first before beginning treatment from day 1 of treatment second after complete treatment after 2 months ,Assessment will be for 5 minutes for ventilatory function
  will be assessed by using Spirometry (smartSOFTmee version 2.14.21)
  FVC (Forced Vital Capacity):
  The maximum volume of air that a person can forcibly exhale after taking a full, deep inhalation. FEV₁ (Forced Expiratory Volume in 1 second):
  The volume of air exhaled during the first second of the forced expiratory maneuver. FEV₁/FVC ratio:
  The percentage of the total forced vital capacity exhaled in the first second, used to assess the presence of airflow obstruction.
  After preparing the device and the patient and delivering instructions, each patient will assume the sitting position with a nose clip on the nose, they will asked to take a deep breath quickly, with a hold of more than one second at TLC, next, firmly seal the mouthpiece with the lips, then execute the FVC technique. Lastly, forcefully exhale for as long as he/she can and as quickly as feasible while loudly asking for more, more, more. This process should last for at least six seconds
Functional capacity by 6MWT | twice ,first before beginning treatment from day 1 of treatment ,second after complete treatment after 2 month Assessment will be for 6 minute
  The 6MWT will be used to measure functional exercise capacity. The investigator measures blood pressure, heart rate, and oxygen saturation. The Patient wears clothing and footwear that are safe for testing. The walking surface will be hard and flat. Often, two cones are set up about 100 feet (30 meters) and the patient will walk back and forth between them for six minutes. At the end of the test, the investigator calculates the distance the patient walked in 6 minutes,

SECONDARY OUTCOMES:
Respiratory muscle strength (MIP and MEP). | twice, first before beginning treatment from day 1 of treatment ,second after complete treatment after 2 month Assessment will be for 3 minute
  it will be used for assessment of respiratory muscle strength. Manometers are pressure reading devices used to measure positive and negative pressures objectively . One manometer developed specifically for maximal expiratory (MEP), and inspiratory (MIP) respiratory pressure testing is the Sonmol Digital Manometer Electric Version.
Patient-reported outcomes by CAT score | twice ,first before beginning treatment from day 1 of treatment ,second after complete treatment after 2 month Assessment will be for 4 minute
  the CAT is a questionnaire that can assess the patient-reported outcomes and the effect of symptoms on COPD patients' lives. The CAT asks eight questions, prompting to assign a score ranging from 0 to 5 for each area A score of 0 means there's no impairment in that area. A score of 5 means severe impairment. The overall score will range from 0 to 40

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin TK, Chen MY, Cheng HH, Chow J, Chen CM, Chou W. Effectiveness of abdominal sandbag training in enhancing diaphragm muscle function and exercise tolerance in patients with chronic respiratory failure. J Formos Med Assoc. 2024 Oct;123(10):1087-1092. doi: 10.1016/j.jfma.2024.01.021. Epub 2024 Feb 1. PMID 38302365
- [Background] • World Health Organization. (2024, November 6). Chronic obstructive pulmonary disease (COPD). Retrieved June 22, 2025, from https://www.who.int/news-room/fact-sheets/detail/chronic-obstructive-pulmonary-disease-(copd)
- [Background] Jing Y, Ma Y, Zhang H, Wu Z, Li Y, Li H, Huang M, Lin L, Xu Y. Pulmonary rehabilitation integrated coached exercise training for patients with COPD: a study protocol for a randomized controlled trial. Trials. 2023 Jan 30;24(1):69. doi: 10.1186/s13063-022-07058-2. PMID 36717916
- [Background] Han B, Chen Z, Ruan B, Chen Y, Lv Y, Li C, Yu L. Effects of Inspiratory Muscle Training in People with Chronic Obstructive Pulmonary Disease: A Systematic Review and Meta-Analysis. Life (Basel). 2024 Nov 12;14(11):1470. doi: 10.3390/life14111470. PMID 39598268
- [Background] Furukawa Y, Miyamoto A, Asai K, Tsutsumi M, Hirai K, Ueda T, Toyokura E, Nishimura M, Sato K, Yamada K, Watanabe T, Kawaguchi T. Respiratory Muscle Strength as a Predictor of Exacerbations in Patients With Chronic Obstructive Pulmonary Disease. Respirology. 2025 May;30(5):408-416. doi: 10.1111/resp.70003. Epub 2025 Feb 26. PMID 40009650
- [Background] Flor-Rufino C, Barrachina-Igual J, Perez-Ros P, Pablos-Monzo A, Martinez-Arnau FM. Resistance training of peripheral muscles benefits respiratory parameters in older women with sarcopenia: Randomized controlled trial. Arch Gerontol Geriatr. 2023 Jan;104:104799. doi: 10.1016/j.archger.2022.104799. Epub 2022 Aug 29. PMID 36070636
- [Background] Chen Q, Wu X, Huang Y, Chen L. Internet of Things-Based Home Respiratory Muscle Training for Patients with Chronic Obstructive Pulmonary Disease: A Randomized Clinical Trial. Int J Chron Obstruct Pulmon Dis. 2024 May 22;19:1093-1103. doi: 10.2147/COPD.S454804. eCollection 2024. PMID 38800522
- [Background] Brito SAF, Scianni AA, Silveira BMF, Oliveira ERM, Mateus ME, Faria CDCM. Effects of high-intensity respiratory muscle training on respiratory muscle strength in individuals with Parkinson's disease: Protocol of a randomized clinical trial. PLoS One. 2023 Sep 8;18(9):e0291051. doi: 10.1371/journal.pone.0291051. eCollection 2023. PMID 37682839
- [Background] Barata PI, Crisan AF, Maritescu A, Negrean RA, Rosca O, Bratosin F, Citu C, Oancea C. Evaluating Virtual and Inpatient Pulmonary Rehabilitation Programs for Patients with COPD. J Pers Med. 2022 Oct 25;12(11):1764. doi: 10.3390/jpm12111764. PMID 36573730
- [Background] • Atef Mohamed, N., Abd Elkader Ahmed, M., & Awadeen, L. (2023). Assessment of quality of life for patients with chronic obstructive pulmonary disease in the outpatient clinic at Beni-Suef University Hospital. Egyptian Journal of Health Care, 14(4), 554-577
- [Background] Aburub A, Darabseh MZ, Badran R, Eilayyan O, Shurrab AM, Degens H. The Effects of Digital Health Interventions for Pulmonary Rehabilitation in People with COPD: A Systematic Review of Randomized Controlled Trials. Medicina (Kaunas). 2024 Jun 11;60(6):963. doi: 10.3390/medicina60060963. PMID 38929580
- See also: Related Info — https://goldcopd.org/2025-gold-report/